CLINICAL TRIAL: NCT07374562
Title: Effect of Stellate Ganglion Block Treatment on Long COVID Symptoms: A Single-Blind, Single-Center Randomized Controlled Trial (STAR-CO)
Brief Title: Stellate Ganglion Block for Long COVID Symptoms: A Randomized Controlled Trial
Acronym: STAR-CO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre intégré universitaire de santé et de services sociaux de la Mauricie-et-du-Centre-du-Québec (Other)
Responsible Party: Principal Investigator, Marie-Claude Lehoux, Principal Investigator, Centre intégré universitaire de santé et de services sociaux de la Mauricie-et-du-Centre-du-Québec
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2026-898; 1028 (Registry Identifier: Base de données des projets de recherche du CIUSSS-MCQ)
Record Dates: First submitted 2026-01-21; First posted 2026-01-29 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Long COVID
Keywords: Long COVID; Stellate Ganglion Block; Bupivacaine
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant
Masking Description: The statistician performing the data analysis will also be masked to group assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stellate Ganglion Block with Bupivacaine (Experimental): Participant receives a right-sided stellate ganglion block under ultrasound guidance, using bupivacaine, performed by an anesthesiologist.
  Interventions: Procedure: Stellate Ganglion Block (Bupivacaine)
- Placebo Neck Injection (Placebo Comparator): Participant receives a saline injection into the sternocleidomastoid muscle under the same conditions.
  Interventions: Procedure: placebo saline injection

INTERVENTIONS:
Procedure: Stellate Ganglion Block (Bupivacaine) — A single ultrasound-guided stellate ganglion block is administered on the right side of the neck under sterile conditions by an anesthesiologist. The needle is positioned between the longus colli muscle and the right carotid artery, and 7 mL of 0.5% bupivacaine is injected. Correct placement is verified by ultrasound and confirmed clinically by the expected appearance of Claude Bernard-Horner syndrome following the injection. Participants are observed for approximately 30 minutes after the procedure.
  Arms: Stellate Ganglion Block with Bupivacaine
Procedure: placebo saline injection — A single placebo injection of 6-8 mL of 0.9% normal saline is administered into the right sternocleidomastoid muscle. The procedure uses the same patient positioning, sterile preparation, and ultrasound guidance as the active arm; however, the needle is intentionally placed in the muscle, away from the stellate ganglion, and does not produce a stellate ganglion block (i.e., cannot cause Claude Bernard-Horner syndrome).
  Arms: Placebo Neck Injection

SUMMARY:
This single-center, randomized, controlled, single-blind clinical trial evaluates whether a stellate ganglion block (SGB) using bupivacaine can improve persistent symptoms in adults with long COVID. Participants are assigned in a 1:1 ratio to receive either an ultrasound-guided right-sided SGB or a placebo saline injection delivered to the sternocleidomastoid muscle. After the intervention, participants are followed for 26 weeks with scheduled evaluations that include symptom questionnaires and functional tests.

The study assesses changes in functional status, fatigue, cognitive complaints, quality of life, dyspnea, lower-limb endurance, and orthostatic tolerance over time. Safety is monitored throughout all follow-up visits. Approximately 40 participants meeting predefined eligibility criteria will be enrolled. This trial seeks to determine whether a single stellate ganglion block has an effect on persistent long-COVID symptoms compared with placebo.The results will help determine the therapeutic value of SGB in the management of long COVID and inform future research and clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years and older
* Positive COVID-19 test confirmed by RT-PCR, antibody test, or antigen test at least 3 months prior to randomization, OR presumed COVID-19 evaluated by the site investigator (no positive test required) with an acute illness occurring after October 15, 2019 and at least 3 months prior to randomization.
* Persistent symptoms ≥12 weeks after onset of acute COVID-19 AND symptoms lasting at least 2 months. The onset date is defined as the earliest of: date of first positive test, date of first symptoms
* Post-COVID Functional Status Scale score ≥2.
* Persistent dyspnea ≥2/4 on the mMRC scale at least 12 weeks post-infection.
* Persistent COVID-19-related symptoms at the time of randomization.
* If taking medications for fatigue or cognition (e.g., sildenafil, modafinil, armodafinil, guanfacine, N-acetylcysteine, stimulants for ADHD), these must have been initiated and stable for ≥4 weeks prior to randomization. Participants are asked not to stop or alter these medications during the study if possible.
* Able and willing to provide written informed consent.
* Able to read and understand French.

Exclusion Criteria:

* Prior diagnosis of myalgic encephalomyelitis (ME) or fibromyalgia
* Being on sick leave or disability at the time of the original acute COVID-19 infection.
* Pregnancy or breastfeeding.
* Myocardial infarction within the last 12 weeks.
* Use of anticoagulant therapy.
* Glaucoma.
* Emphysema requiring home oxygen.
* Cardiac conduction abnormalities.
* Known hypersensitivity to bupivacaine.
* Previous stellate ganglion block (SGB) procedure.
* Any condition that, in the judgment of the medical investigator, makes the patient not a candidate for the proposed treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-02-05 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Post-COVID-19 Functional Status Scale (PCFS) | 4 weeks after the intervention
  The PCFS measures limitations in daily functioning related to persistent post-COVID-19 symptoms. Scores range from 0 (no functional limitation) to 4 (severe functional limitation). Assesses changes in functional status over time.
Fatigue Severity Scale (FSS) | 4 weeks after the intervention
  The FSS is a validated 9-item questionnaire assessing the impact of fatigue on daily activities, motivation, and functioning. Each item is scored from 1 to 7; higher scores indicate greater fatigue severity. Clinically significant change is defined as ≥0.45 points.
Brain Fog Scale (BFS) | 4 weeks after the intervention
  The BFS is a 23-item questionnaire evaluating cognitive symptoms associated with Long COVID, including mental fatigue, cognitive clarity, logical thinking, and concentration. Total scores range from 0 to 92, with higher scores indicating more severe cognitive impairment.

SECONDARY OUTCOMES:
Health-Related Quality of Life (SF-36) | 4 weeks after the intervention
  The SF-36 is a validated 36-item questionnaire assessing eight domains of health-related quality of life, including physical functioning, limitations due to physical or emotional problems, pain, general health, vitality, social functioning, and mental health. Higher scores reflect better perceived health and functioning.
Dyspnea Severity (mMRC Scale) | 4 weeks after the intervention
  The modified Medical Research Council (mMRC) Dyspnea Scale is a 0-4 grading system that assesses the degree to which breathlessness limits daily activities. Higher grades indicate greater functional limitation due to dyspnea. It is the only validated French-language scale measuring dyspnea in daily activities.
Lower-Limb Muscle Endurance (1-Minute Sit-to-Stand Test) | 4 weeks after the intervention
  The 1-Minute Sit-to-Stand Test (1STST) measures lower-limb muscular endurance by counting the number of sit-to-stand repetitions a participant completes in one minute from a standard chair without armrests. It is reliable, sensitive, and well-tolerated in populations with impaired physical capacity. Higher counts indicate better endurance.
Orthostatic Intolerance (NASA Lean Test) | 4 weeks after the intervention
  The NASA Lean Test assesses orthostatic intolerance by measuring heart rate and blood pressure changes during 10 minutes of standing with the back supported against a wall. Results help identify symptoms such as dizziness, palpitations, or light-headedness related to positional changes. If a participant cannot complete 10 minutes, the test is still considered valid.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre hospitalier affilié universitaire régional, Trois-Rivières, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided